CLINICAL TRIAL: NCT00489281
Title: A Phase II Trial of Non-Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched and HLA-Matched Bone Marrow for Patients With Sickle Cell Anemia and Other Hemoglobinopathies
Brief Title: Non-Myeloablative Bone Marrow Transplant for Patients With Sickle Cell Anemia and Other Blood Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Initiation of CMS BMT study for sickle-cell disease operating under NCT01166009 made further accrual to this study impossible.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0676; P30CA006973 (NIH); P01CA015396 (NIH); NA_00002479 (Other: JHMIRB)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Mycophenolic Acid; Sirolimus; Levetiracetam; Antilymphocyte Serum; thymoglobulin

ARMS (2):
- Transplant - 200 cGy (Experimental): Conditioning regimen with anti-thymocyte globulin, fludarabine, cyclophosphamide, and total body irradiation - 200. Seizure prophylaxis with levetiracetam. Allogeneic bone marrow transplant infusion on Day 0. Graft-vs-host-disease (GVHD) prophylaxis with cyclophosphamide, mycophenolate mofetil, and sirolimus.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mycophenolate mofetil; Drug: Sirolimus; Procedure: Allogeneic bone marrow transplant; Radiation: Total body irradiation - 200; Drug: Levetiracetam; Biological: Anti-thymocyte globulin
- Transplant - 400 cGy (Experimental): Conditioning regimen with anti-thymocyte globulin, fludarabine, cyclophosphamide, and total body irradiation - 400. Seizure prophylaxis with levetiracetam. Allogeneic bone marrow transplant infusion on Day 0. Graft-vs-host-disease (GVHD) prophylaxis with cyclophosphamide, mycophenolate mofetil, and sirolimus.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mycophenolate mofetil; Drug: Sirolimus; Procedure: Allogeneic bone marrow transplant; Drug: Levetiracetam; Biological: Anti-thymocyte globulin; Radiation: Total body irradiation - 400

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (Cy) 14.5 mg/kg/day intravenously (IV) on Days -6 and -5 and 50 mg/kg/day IV on Days +3 and +4.
  Other Names: Cytoxan; Cy; CTX
Drug: Fludarabine — Fludarabine 30 mg/m^2/day IV on Days -6, -5, -4, -3, and -2.
  Other Names: Fludara
Drug: Mycophenolate mofetil — Mycophenolate mofetil 15 mg/kg by mouth (PO) three times a day from Day +5 to Day +35.
  Other Names: MMF; CellCept
Drug: Sirolimus — The first dose of Sirolimus is 6 mg PO on Day +5. Further dosing is adjusted according to drug levels. Sirolimus is continued through Day +365.
  Other Names: Rapamune
Procedure: Allogeneic bone marrow transplant — An allogeneic bone marrow transplant is a procedure that involves taking bone marrow from a donor and giving it to a recipient.
  Other Names: Allo BMT
Radiation: Total body irradiation - 200 — 200 centigray (cGy) in one fraction on Day -1.
  Other Names: TBI
  Arms: Transplant - 200 cGy
Drug: Levetiracetam — Given at 500 mg PO twice daily from Day -6 to Day +365.
  Other Names: Keppra
Biological: Anti-thymocyte globulin — Test dose of 0.5 mg/kg IV given on Day -9, then 2 mg/kg/day IV on Day -8 and -7.
  Other Names: ATG; Thymoglobulin
Radiation: Total body irradiation - 400 — 400 centigray (cGy) in one fraction on Day -1.
  Other Names: TBI
  Arms: Transplant - 400 cGy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and cyclophosphamide, and total-body irradiation before a donor bone marrow transplant helps stop the growth of abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving sirolimus and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation followed by a donor bone marrow transplant works in treating patients with sickle cell anemia and other blood disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the transplant-related mortality and progression-free survival of patients with severe hemoglobinopathies receiving nonmyeloablative conditioning comprising fludarabine phosphate, cyclophosphamide, and total-body irradiation followed by partially HLA-mismatched bone marrow transplantation from first-degree relatives or HLA-matched donors.
* Characterize donor hematopoietic chimerism at 30, 60, and 180 days after transplantation in these patients.
* Determine the hematologic and non-hematologic toxicity of this regimen in these patients.

OUTLINE:

* Preparative regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1-2 hours on days -6 and -5. Patients also undergo total-body irradiation on day -1.
* Bone marrow transplantation: Patients undergo allogeneic bone marrow transplantation on day 0. Patients then receive cyclophosphamide IV over 1-2 hours on days 3 and 4.
* Graft-versus-host disease prophylaxis: Patients receive sirolimus orally daily on days 5-365 and oral mycophenolate mofetil 3 times a day on days 5-35.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following sickle cell anemias (Hb SS):

  * Hb S/β° thalassemia
  * Hb S/β+ thalassemia
  * Hb SC disease
  * Hb SE disease
  * Hb SD disease
  * Hemoglobin SO-Arab disease
  * Hb S/hereditary persistence of fetal hemoglobin
* Meets 1 of the following criteria:

  * History of invasive pneumococcal disease
  * Stroke or CNS event lasting > 24 hours
  * MRI changes indicative of brain parenchymal damage
  * Evidence of cerebrovascular disease by magnetic resonance angiography
  * Acute chest syndrome requiring exchange transfusion or hospitalization
  * Recurrent vaso-occlusive pain crisis (> 2 per year for the last 2 years)
  * Stage I or II sickle lung disease
  * Sickle retinopathy
  * Osteonecrosis
  * Red cell alloimmunization (> 2 antibodies) during long-term transfusion
  * Constellation of dactylitis in the first year of life AND a baseline hemoglobin < 7 g/dL and leukocytosis (WBC > 13.4/mm^3) in the absence of infection during the second year of life
  * Pitted RBC count > 3.5% during the first year of life
* Ineligible for or refused bone marrow transplantation from an HLA-matched sibling donor
* Partially mismatched (at least haploidentical) first-degree relative donor available

  * No minor (donor anti-recipient) ABO incompatibility if an ABO compatible donor is available

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky or Lansky PS 70-100%
* LVEF ≥ 35%
* FEV_1 and forced vital capacity ≥ 40% predicted
* Direct bilirubin < 3.1 mg/dL
* No moderate to severe pulmonary hypertension by ECHO
* No debilitating medical or psychiatric illness that would preclude study participation
* No HIV positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior transfusions from donor
* No immunosuppressive agents, including steroids as antiemetics, within 24 hours after the last dose of post-transplantation cyclophosphamide

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-06-23 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bolanos-Meade, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldenberg M, Varadhan R, Gamper CJ, Cooke KR, Ambinder AJ, Symons HJ, Pecker LH, Jones RJ, Brodsky RA, Bolanos-Meade J. Bone marrow transplantation for sickle cell disease using post-transplantation cyclophosphamide and 400 cGy TBI. Blood Adv. 2026 Jan 22:bloodadvances.2025017413. doi: 10.1182/bloodadvances.2025017413. Online ahead of print. PMID 41569644
- [Derived] Bolanos-Meade J, Cooke KR, Gamper CJ, Ali SA, Ambinder RF, Borrello IM, Fuchs EJ, Gladstone DE, Gocke CB, Huff CA, Luznik L, Swinnen LJ, Symons HJ, Terezakis SA, Wagner-Johnston N, Jones RJ, Brodsky RA. Effect of increased dose of total body irradiation on graft failure associated with HLA-haploidentical transplantation in patients with severe haemoglobinopathies: a prospective clinical trial. Lancet Haematol. 2019 Apr;6(4):e183-e193. doi: 10.1016/S2352-3026(19)30031-6. Epub 2019 Mar 14. PMID 30878319

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was a screen failure.
Period: Overall Study
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
Started | 29 | 13
Completed | 29 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy | Total
Number analyzed (Participants) | 29 | 13 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 6 | 15
  Between 18 and 65 years | 20 | 7 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 19 [6 to 42] | 21 [5 to 31] | 21 [5 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 12 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 13 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 6 | 31
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 13 | 42
Disease [Count of Participants; unit: Participants]
  Sickle cell disease | 25 | 7 | 32
  Thalassemia | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Transplant-related Mortality
Description: Number of participants who died for reasons related to bone marrow transplant.
Time Frame: Up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
Number analyzed (Participants) | 29 | 13
Participants | 1 | 0

2. Primary Outcome: Progression-free Survival
Description: Percentage of participants who are alive without relapse.
Time Frame: 2 years
Population: Due to early study termination, data was not collected to assess this outcome measure
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Donor Chimerism at 30 Days
Description: Number of participants with full (95-100%), mixed (5-94%), and no (0-4%) donor cells. Chimerism is reported for unsorted whole blood and T cells.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
Number analyzed (Participants) | 29 | 13
Participants
  Whole blood: 95-100% | 12 | 8
  Whole blood: 5-94% | 15 | 3
  Whole blood: 0-4% | 1 | 1
  Whole blood: Unknown or not measured | 1 | 1
  T cells: 95-100% | 4 | 4
  T cells: 5-94% | 18 | 8
  T cells: 0-4% | 5 | 0
  T cells: Unknown or not measured | 2 | 1

4. Secondary Outcome: Donor Chimerism at 1 Year
Description: as for outcome 3
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
Number analyzed (Participants) | 29 | 13
Participants
  Whole blood: 95-100% | 6 | 9
  Whole blood: 5-94% | 9 | 3
  Whole blood: 0-4% | 1 | 0
  Whole blood: Unknown or not measured | 13 | 1
  T cells: 95-100% | 7 | 10
  T cells: 5-94% | 9 | 2
  T cells: 0-4% | 0 | 0
  T cells: Unknown or not measured | 13 | 1

ADVERSE EVENTS:
Time Frame: Up to 60 days
Description: Only serious adverse events and grade 3-5 non-serious adverse events were collected.
Arm/Group | Transplant - 200 cGy | Transplant - 400 cGy
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/13
Serious Adverse Events (participants affected / at risk) | 21/29 | 7/13
Other Adverse Events (participants affected / at risk) | 0/29 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant - 200 cGy (N=29) | Transplant - 400 cGy (N=13)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 4 (4) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Central line thrombosis (Vascular disorders) | 1 (1) | 0 (0)
CLABSI (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 4 (6) | 0 (0)
Hallucination (Nervous system disorders) | 1 (2) | 0 (0)
Headache (General disorders) | 4 (4) | 1 (1)
Hematoma (General disorders) | 1 (1) | 0 (0)
Herpes simplex virus (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalemia (Investigations) | 1 (1) | 0 (0)
Influenza A (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 8 (8) | 5 (6)
Pain - abdomen (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pain - ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - back (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Pain - bone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - chest (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain - flank (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - unspecified (General disorders) | 3 (4) | 0 (0)
Vaso-occlusive crisis (Blood and lymphatic system disorders) | 10 (22) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 4 (4) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory syncytial virus (Infections and infestations) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT00489281/Prot_SAP_000.pdf